CLINICAL TRIAL: NCT00794001
Title: Feedback Intervention and Treatment Times in ST- Elevation Myocardial Infarction (FITT-STEMI): A Multicenter Trial Analyzing the Effects of Systematic Data Feedback on Treatment Quality and Survival Rates.
Brief Title: Feedback Intervention and Treatment Times in ST- Elevation Myocardial Infarction
Acronym: FITT-STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Heinrich Scholz (Other)
Collaborators: ALKK: Arbeitsgemeinschaft Leitender Kardiologischer Krankenhausaerzte (Unknown); The German Heart Foundation (Other); Aerztekammer Niedersachsen (Unknown)
Responsible Party: Sponsor-Investigator, Karl Heinrich Scholz, Professor Dr., St.Bernward Hospital
Organization: St.Bernward Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GOE-01-10-07
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; angioplasty; data feedback; continuous quality improvement; STEMI; Feedback; Quality Assurance, Health Care; Emergency service hospital
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Data Feedback (Experimental): The intervention is systematic feedback on performance (using predefined quality indicators) to cardiology, ED, and EMS-stakeholders and staff.
  Interventions: Behavioral: Data analysis and Feedback

INTERVENTIONS:
Behavioral: Data analysis and Feedback — Data analysis feedback: quarterly meetings with all stakeholders to present data and discuss potential areas of improvement.

SUMMARY:
Part I (Pilot Phase): The purpose of this study is to examine if formalized data assessment and systematic feedback improves treatment times (i.e. contact-to-balloon time and door-to-balloon time) in patients with myocardial infarction with ST-segment elevation (STEMI).

Part II (Implementation Phase): The Purpose is to prospectively investigate if survival can be improved by stringent use of this concept of formalized data analysis and systematic feedback of procedural and clinical data to all participating physicians and other members of the STEMI patients treating personnel.

Part III (Advance Phase): The purpose is to develop, introduce and evaluate prospectively an automated, highly standardized feedback tool informing participating centers on key performance characteristics (procedural and clinical outcomes).

DETAILED DESCRIPTION:
For many patients with myocardial infarction with ST-segment elevation (STEMI), the time from presentation to percutaneous coronary intervention (PCI) exceeds established goals. Formalized data feedback is one strategy proposed to reduce treatment time in STEMI-patients. The aim of this multicenter study is to evaluate whether systematic data analysis and feedback leads to shorter contact-to-balloon and door-to-balloon times and reduces mortality in different regional care networks serving patients with STEMI. The multicenter trial includes hospitals with primary percutaneous coronary intervention (PCI) capacity. Existing protocols encourage prompt transfer of patients with STEMI to the PCI center and emphasize minimizing time to treatment. In each participating center, all patients presenting with STEMI are enrolled. The study is conducted prospectively during five consecutive 3-month periods (quarters). Data collection is web-based and identical for the five quarters. For each center, time points from initial contact with the medical system to revascularization are assessed, analyzed and presented in an interactive session to hospital and emergency services staff. This formalized data feedback is performed at the end of each quarter.

The multi-phase FITT-STEMI project is structured as follows:

Part I (Pilot Phase)

Patients presenting during the first three-month period are included as the reference group. Data from patients with STEMI presenting during the next four quarters are presented in the same manner. Comparisons between the reference group and the next quarters will be made with the Gehan and Pearson χ2 tests.

Part II (Implementation Phase)

Following the Pilot Phase started as feasibility study including a group of 6 different hospital systems of STEMI care, the multicenter FITT-STEMI-Implementation-Phase was started to investigate the effect of standardized documentation, analysis and systematic feedback-intervention on prognosis within a large group of different hospitals capable of primary PCI. This study is performed over 6 quarters including 3 feedback-sessions, and so far, 46 different PCI-hospitals capable of primary PCI participate at the FITT-STEMI-implementation-phase.

Following the initial study period with quarterly feedback-sessions, data collection is continued, and in all of these hospitals feedback-sessions with the EMS- and hospital-staff are held once a year (after quarters 8, 12, 16, and so on).

Participating hospitals So far, a total of 53 hospital-systems with primary PCI capacity and cooperating non-PCI-hospitals participate at the FITT-STEMI-program. At the PCI-Centers, 24 h PCI capability existing for at least one year prior to inclusion, at least two interventional cardiologists who could take call, and a volume of at least 250 PCI procedures as well as 50 PCI procedures in STEMI patients per year are required for participation at the project. All 6 key strategies of the ACC D2B-initiative (Bradley EH, NEJ 2006) were endorsed by the hospitals before participating in the project. All hospitals ensured prompt transfer of patients with STEMI to the PCI centers minimizing time to treatment.

The overall geographic catchment area currently serves a population of more than 10 million people in Germany with more than 5,500 STEMI patients per year, which is consistent with > 10 % of the German population and with > 10% of the patients treated with acute STEMI in German hospitals per year. Estimated Enrollment: 50,000 participants (Phases I and II).

Part III (Advance Phase)

This phase of the multi-phase FITT-STEMI aims to develop, introduce and evaluate prospectively an automated, highly standardized feedback tool informing participating centers on key performance characteristics (procedural and clinical outcomes). A stepped wedge design with baseline phase will be used. The participating (newly recruited or already established) centres will be randomly allocated to switching over from the implemented feedback form to the new automated, highly standardized feedback tool; the switch-over process is staggered over time. Estimated Enrollment: 60,000 participants (Phases I - III).

ELIGIBILITY:
Inclusion Criteria:

* all patients who received a diagnosis of STEMI* and were transported to the cardiac catheterization laboratory of the primary PCI center with the intention to perform primary PCI.

  * STEMI definition:
* elevation of the ST-segments of greater than or equal to 0.1 mV in at least two contiguous limb- or precordial leads
* new or presumable new left bundle branch block in the presence of typical symptoms

Exclusion Criteria:

* STEMI-patients with duration of infarct-related symptoms longer than 24 hours are excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2007-10; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Contact to Balloon Time | six consecutive three month periods (quarters)

SECONDARY OUTCOMES:
mortality (in-hospital-mortality; 30-day-mortality; 1-year-mortality) | six consecutive three month periods (quarters)

CONTACTS AND LOCATIONS:
Overall Officials: Karl H. Scholz, MD., Study Director — St.Bernward Hospital
Locations (1):
- St.Bernward Hospital, Hildesheim, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ting HH, Krumholz HM, Bradley EH, Cone DC, Curtis JP, Drew BJ, Field JM, French WJ, Gibler WB, Goff DC, Jacobs AK, Nallamothu BK, O'Connor RE, Schuur JD; American Heart Association Interdisciplinary Council on Quality of Care and Outcomes Research, Emergency Cardiovascular Care Committee; American Heart Association Council on Cardiovascular Nursing; American Heart Association Council on Clinical Cardiology. Implementation and integration of prehospital ECGs into systems of care for acute coronary syndrome: a scientific statement from the American Heart Association Interdisciplinary Council on Quality of Care and Outcomes Research, Emergency Cardiovascular Care Committee, Council on Cardiovascular Nursing, and Council on Clinical Cardiology. Circulation. 2008 Sep 2;118(10):1066-79. doi: 10.1161/CIRCULATIONAHA.108.190402. Epub 2008 Aug 13. No abstract available. PMID 18703464
- [Result] Scholz KH, Hilgers R, Ahlersmann D, Duwald H, Nitsche R, von Knobelsdorff G, Volger B, Moller K, Keating FK. Contact-to-balloon time and door-to-balloon time after initiation of a formalized data feedback in patients with acute ST-elevation myocardial infarction. Am J Cardiol. 2008 Jan 1;101(1):46-52. doi: 10.1016/j.amjcard.2007.07.078. Epub 2007 Nov 19. PMID 18157964
- [Result] Scholz KH, von Knobelsdorff G, Ahlersmann D, Keating FK, Jung J, Werner GS, Nitsche R, Duwald H, Hilgers R. [Optimizing systems of care for patients with acute myocardial infarction. STEMI networks, telemetry ECG, and standardized quality improvement with systematic data feedback]. Herz. 2008 Mar;33(2):102-9. doi: 10.1007/s00059-008-3120-6. German. PMID 18344028
- [Result] Scholz KH, Maier SK, Jung J, Fleischmann C, Werner GS, Olbrich HG, Ahlersmann D, Keating FK, Jacobshagen C, Moehlis H, Hilgers R, Maier LS. Reduction in treatment times through formalized data feedback: results from a prospective multicenter study of ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2012 Aug;5(8):848-57. doi: 10.1016/j.jcin.2012.04.012. PMID 22917457
- [Result] Maier LS, Maier SK, Scholz KH. Letter by Maier et al regarding article, "Emergency department bypass for ST-segment-elevation myocardial infarction patients identified with a prehospital electrocardiogram: a report from the American Heart Association Mission: Lifeline Program". Circulation. 2014 Mar 4;129(9):e371. doi: 10.1161/CIRCULATIONAHA.113.005631. No abstract available. PMID 24589702
- [Result] Scholz KH, Maier SKG, Maier LS, Lengenfelder B, Jacobshagen C, Jung J, Fleischmann C, Werner GS, Olbrich HG, Ott R, Mudra H, Seidl K, Schulze PC, Weiss C, Haimerl J, Friede T, Meyer T. Impact of treatment delay on mortality in ST-segment elevation myocardial infarction (STEMI) patients presenting with and without haemodynamic instability: results from the German prospective, multicentre FITT-STEMI trial. Eur Heart J. 2018 Apr 1;39(13):1065-1074. doi: 10.1093/eurheartj/ehy004. PMID 29452351
- [Result] Scholz KH, Friede T, Meyer T, Jacobshagen C, Lengenfelder B, Jung J, Fleischmann C, Moehlis H, Olbrich HG, Ott R, Elsasser A, Schroder S, Thilo C, Raut W, Franke A, Maier LS, Maier SK. Prognostic significance of emergency department bypass in stable and unstable patients with ST-segment elevation myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2020 Mar;9(1_suppl):34-44. doi: 10.1177/2048872618813907. Epub 2018 Nov 27. PMID 30477317
- [Result] Scholz KH, Lengenfelder B, Jacobshagen C, Fleischmann C, Moehlis H, Olbrich HG, Jung J, Maier LS, Maier SK, Bestehorn K, Friede T, Meyer T. Long-term effects of a standardized feedback-driven quality improvement program for timely reperfusion therapy in regional STEMI care networks. Eur Heart J Acute Cardiovasc Care. 2021 May 25;10(4):397-405. doi: 10.1177/2048872620907323. Epub 2020 Jul 29. PMID 32723177
- [Result] Scholz KH, Lengenfelder B, Thilo C, Jeron A, Stefanow S, Janssens U, Bauersachs J, Schulze PC, Winter KD, Schroder J, Vom Dahl J, von Beckerath N, Seidl K, Friede T, Meyer T. Impact of COVID-19 outbreak on regional STEMI care in Germany. Clin Res Cardiol. 2020 Dec;109(12):1511-1521. doi: 10.1007/s00392-020-01703-z. Epub 2020 Jul 16. PMID 32676681
- [Result] Scholz M, Meyer T, Maier LS, Scholz KH. Infarct-Related Artery as a Donor of Collaterals in ST-Segment-Elevation Myocardial Infarction With Concomitant Chronic Total Occlusion: Challenge of the Double-Jeopardy Thesis. J Am Heart Assoc. 2023 Apr 4;12(7):e028115. doi: 10.1161/JAHA.122.028115. Epub 2023 Mar 21. PMID 36942757
- [Derived] Scholz P, Friede T, Scholz KH, Grabmaier U, Meyer T, Seidler T. Pre-hospital heparin is not associated with infarct vessel patency and mortality in ST-segment elevation myocardial infarction patients with out-of-hospital cardiac arrest. Clin Res Cardiol. 2024 Aug 1. doi: 10.1007/s00392-024-02499-y. Online ahead of print. PMID 39088062
- [Derived] Scholz KH, Meyer T, Lengenfelder B, Vahlhaus C, Tongers J, Schnupp S, Burckhard R, von Beckerath N, Grusnick HM, Jeron A, Winter KD, Maier SKG, Danner M, Vom Dahl J, Neef S, Stefanow S, Friede T. Patient delay and benefit of timely reperfusion in ST-segment elevation myocardial infarction. Open Heart. 2021 May;8(1):e001650. doi: 10.1136/openhrt-2021-001650. PMID 33958491
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/18157964?ordinalpos=3&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum